CLINICAL TRIAL: NCT03101189
Title: A Single-center, Double-blind, Placebo-controlled, Randomized Study to Investigate the Tolerability, Safety, Pharmacokinetics, and Pharmacodynamics of Single- and Multiple-dose ACT-541468 in Healthy Japanese and Caucasian Subjects
Brief Title: A Study of ACT-541468 in Healthy Japanese and Caucasian Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: AC-078-105
Record Dates: First submitted 2017-03-24; First posted 2017-04-05 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Healthy Subjects
Keywords: safety; Japanese; pharmacokinetics
MeSH Terms: interventions — daridorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ACT-541468 (25 mg) (Experimental): 8 Japanese and 8 Caucasian subjects will receive 25 mg (1 capsule) of ACT-541468 once daily for 5 days
  Interventions: Drug: ACT-541468
- ACT-541468 (50 mg) (Experimental): 8 Japanese and 8 Caucasian subjects will receive 50 mg (2 capsules) of ACT-541468 once daily for 5 days
  Interventions: Drug: ACT-541468
- Placebo (Placebo Comparator): 2 Japanese / 2 Caucasian subjects will receive 1 placebo capsule to match subjects in the ACT-541468 (25 mg) group and 2 other Japanese / 2 Caucasian subjects will receive 2 placebo capsules to match subjects in the ACT-541468 (50 mg) group
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ACT-541468 — Capsule
  Arms: ACT-541468 (25 mg); ACT-541468 (50 mg)
Drug: placebo — Matching placebo capsule
  Arms: Placebo

SUMMARY:
So far, ACT-541468 has been studied mainly in Caucasian subjects. The present study will bridge results obtained in Caucasian subjects to those in Japanese subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent form;
* Healthy male and female subjects aged between 20 and 50 years (inclusive) at screening;
* Negative serum pregnancy tests at screening and negative urine pregnancy test at Day 1 for women of childbearing potential and agreement to use a reliable method of contraception for at least 90 days after last study drug intake;
* Body mass index (BMI) of 18.0 to 26.0 kg/m2 (inclusive) at screening;
* Healthy on the basis of physical examination, cardiovascular assessments and laboratory tests;
* Caucasian or Japanese ethnicity.

Japanese subjects only:

* must be of native Japanese descent (all parents/grandparents of Japanese descent);
* must not have been away from Japan for more than 10 years (at screening visit);
* lifestyle should not have changed significantly since relocation from Japan.

Key Exclusion Criteria:

* Any contraindication to the study treatments;
* History or clinical evidence of any disease or medical / surgical condition or treatment, which may put the subject at risk of participation in the study or may interfere with the absorption, distribution, metabolism or excretion of the study treatments;
* History of narcolepsy or cataplexy or modified Swiss narcolepsy scale total score < 0;
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-04-24 (Actual); Study Completion 2017-04-26 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of ACT-541468 | From Day1 pre-dose to 48 hours after the last dose on Day 5
  The geometric mean Cmax values will be calculated based on pharmacokinetic (PK) blood sampling
Area under the plasma concentration-time curves during a dosing interval [AUC(0-24)] of ACT-541468 | From Day1 pre-dose to 48 hours after the last dose on Day 5
  The geometric mean AUC(0-24) values will be calculated based on PK blood sampling

SECONDARY OUTCOMES:
Time to reach Cmax (tmax) of ACT-541468 | From Day1 pre-dose to 48 hours after the last dose on Day 5
  The median tmax values will be calculated based on PK blood sampling
Terminal half-life [t(1/2)] of ACT-541468 | From Day1 pre-dose to 48 hours after the last dose on Day 5
  The geometric mean t(1/2) values will be calculated based on PK blood sampling
Area under the plasma concentration-time curves from time 0 to 8 h [AUC(0-8)] | From Day1 pre-dose to 48 hours after the last dose on Day 5
  The geometric mean AUC(0-8) values will be calculated based on PK blood sampling
Incidence of treatment-emergent adverse events | Up to Day 7 (end of study)
  The percentage of subjects with treatment-emergent adverse events will be reported
Incidence of adverse events leading to premature discontinuation of study treatment | Up to Day 5
  The number of subjects who prematurely discontinued the study treatment due to an adverse event will be reported
Incidence of any clinical relevant findings in ECG variables | Up to Day 7 (end of study)
  The number of subjects with any treatment-emergent electrocardiogram (ECG) abnormalities will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Muehlan, Study Director — Actelion
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No